CLINICAL TRIAL: NCT03843801
Title: A Prospective Study to Evaluate the Suture Pattern With the Endomina Suturing Device for Endoscopic Sutured Gastroplasty (ESG).
Acronym: Pattern
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCB : / B406201838475
Record Dates: First submitted 2019-02-14; First posted 2019-02-18 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Obesity
Keywords: Endoscopy; Mini invasive
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Volume reduction (Active Comparator): Intragastric sutures are done to reduce the volume of the stomach
  Interventions: Device: Endomina
- Gastric emptying reduction (Active Comparator): Intragastric sutures are done to slower the gastric emptying
  Interventions: Device: Endomina
- Increasing distension (Active Comparator): Intragastric sutures are done to maximalize the gastric distension
  Interventions: Device: Endomina

INTERVENTIONS:
Device: Endomina — The intervention will be performed under general anesthesia with tracheal intubation. Endomina will be introduced into the stomach over guide wires and then fixed to the endoscope. The procedure will include the placement of transmural anterior-posterior sutures in the stomach in order to achieve a gastric remodelling. Patient will be kept overnight after the procedure.

SUMMARY:
Advances in endoluminal devices are now allowing clinicians the ability to begin exploring bariatric procedures performed via flexible endoscopy. Although these procedures may not be as effective as their surgical counterparts, these less-invasive options may relieve patients of the significant risks associated with surgery (1).

Endomina (Endo Tools Therapeutics, Gosselies, Belgium) is CE mark device that may be attached to an endoscope inside the body and allows remote manipulation of the arms of the device during a peroral intervention. It offers the possibilities of making transoral surgical full thickness sutures and may allow performing endoscopic therapeutic interventions, via a transoral route.

A first trial including 11 patients assessed feasibility and safety of the technique (2). There were no complications and the short-term results were encouraging. Then a multicentric efficacy study was conducted, including 51 patients (3). The results where EWL of 31% at one year and TBWL of 9% without complications.

Finally a randomized controlled study was done including 73 patients in a 2/1 randomized fashion with a crossover at 6 months. Treated group was with the endomina device and controlled group was diet only. The follow-up was the same in each group. Primary endpoint was to reach the ASGE guideline "difference between a control group and a treatment group of minimum 15%" (4).

Technique and suture pattern have evolved since the first study. The aim of this prospective evaluation is to compare different suture patterns and their mechanism of action.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-64 years;
2. BMI between 30 to 40 kg/m²
3. Must be able to comply with all study requirements for the duration of the study as outlined in the protocol. This includes complying with the visit schedule as well as study specific procedures such as: clinical assessment, endoscopy, radiography, gastric emptying scintigraphy, satiety test, as well as laboratory investigations.
4. Must be able to understand and be willing to provide written informed consent.
5. Must have completed the multidisciplinary workup

Exclusion Criteria:

1. Achalasia and any other esophageal motility disorders
2. Heart diseases: unstable angina, myocardial infarction within the past year, or heart disease classified within the New York Heart Association's Class III or IV functional capacity.
3. Hypertension: uncontrolled hypertension during last 3 month
4. Severe renal, hepatic, pulmonary disease or cancer;
5. GI stenosis or obstruction
6. Pregnancy or breastfeeding or willing to become pregnant within study duration
7. History of gastric surgery (any type)
8. Impending gastric surgery 60 days post intervention
9. History of weight changes (±5% TBWL) within the previous 6 months
10. Placement/removal of an intragastric balloon in less than 6 months
11. Currently participating in other study
12. HP positive

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2020-11-26 (Actual); Study Completion 2020-11-26 (Actual)

PRIMARY OUTCOMES:
Weight loss | one year from procedure
  no difference in weight loss between groups

SECONDARY OUTCOMES:
Gastric emptying | one year from procedure
  Evaluation of the correlation between gastric emptying scintigraphy results and the suture pattern related to motility disruption
Satiety test assessed by the correlation between satiety test and the suture pattern related to volume reduction | one year from procedure
  Evaluation of the correlation between satiety test and the suture pattern related to volume reduction
sutures | one year from procedure
  Evaluation of the correlation between the number of remaining sutures (with gastric remodeling) and weight loss
Excess weight loss | one year from procedure
  Percentage of patients, total and per group, reaching ASGE guidelines of 25% Excess weight loss at 1-year

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - CUB Hopital erasme, Anderlecht
  - Gastroenterology Department Erasme Hospital, Brussels

IPD SHARING:
Plan to Share IPD: No